CLINICAL TRIAL: NCT02419781
Title: Recovery by Endovascular Salvage for Cerebral Ultra-acute Embolism (RESCUE)-Japan Randomized Controlled Trial
Brief Title: Recovery by Endovascular Salvage for Cerebral Ultra-acute Embolism (RESCUE)-Japan RCT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Evidence of thrombectomy for acute stroke was established
Sponsor: Shinichi Yoshimura (Other)
Responsible Party: Sponsor-Investigator, Shinichi Yoshimura, Professor, Hyogo Medical University
Organization: Hyogo Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMIN000015272
Record Dates: First submitted 2015-01-19; First posted 2015-04-17 (Estimated); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group with endovascular treatment (Active Comparator): Group with additional endovascular treatment
  Interventions: Procedure: Rescue endovascular therapy
- Group without endovascular treatment (Active Comparator): Group without additional endovascular treatment
  Interventions: Procedure: No endovascular therapy

INTERVENTIONS:
Procedure: Rescue endovascular therapy — endovascular treatment using any devises for acute ischemic stroke patients with large vessel occlusion and not respond to intravenous recombinant tissue plasminogen activator (rt-PA) therapy
  Arms: Group with endovascular treatment
Procedure: No endovascular therapy
  Arms: Group without endovascular treatment

SUMMARY:
The aim of this study is to clarify the efficacy of the endovascular treatment for acute ischemic stroke patients with large vessel occlusion and are not respond to intravenous recombinant tissue plasminogen activator (rt-PA) therapy.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke patients who were treated with intravenous rt-PA therapy within 4.5 hours from onset and have persistent occlusion of IC and M1 proximal portion* confirmed by cerebral angiography.

  *: M1 proximal portion means the segment of MCA within 5mm from the internal carotid bifurcation.
* Patients who can receive endovascular treatment within 8 hours after the onset.
* Patients whose DWI-ASPECTS was 5 points and more, or CT-ASPECT was 6 points and more just before cerebral angiography.
* Patients whose NIHSS is between 8 and 29 points.
* Patients who are between 20 and 85 years.
* Gender does not matter.
* Consent of this study participants must be obtained from patients or legal representative in writing.

Exclusion Criteria:

* Patients whose neurological symptoms improved and NIHSS is eight points and less after intravenous rt-PA therapy.
* Patients whose mRS was 3 points and more before the onset. 3)Patients with past history of lumbar puncture or arterial puncture that were difficult of hemostasis.
* Patients with intracranial tumor
* Patients with hypersensitivity to contrast agent.
* Patients with serious renal disease.
* Patients with malignant tumor.
* Patients with pregnancy or suspect of pregnancy, or during lactation.
* Patients with findings of acute myocardial infarction or pericarditis after myocardial infarction.
* Patients who cannot be followed for 3 months.
* Patients with past history of cerebral aneurysm, cerebral arteriovenous malformation, cerebral venous thrombosis, or moyamoya disease.
* Patients with other occlusions besides ICA or M1 proximal portion.
* Patients with aortic dissection complicating endovascular treatment.
* Patients with tortuous arteries that prevent the navigation of the device to the target vessel.
* Patients considered inappropriate to participate in the study.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-10; Primary Completion 2017-03 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Assessment of modified Rankin Scale shift analysis at 90 days after onset | 90 days

SECONDARY OUTCOMES:
The rate of mRS 0-2 at 90 days (+/- 10 days) after onset | 90 days
Death within 90 days (+/- 10 days) after onset | 90 days
Revascularization rates of the target vessel at 72 hours (+/- 8 hours) after onset | 72 hours
  for CT angiography or MR angiography
Symptomatic intracranial hemorrhage within 72 hours (+/- 8 hours) after onset | 72 hours
The difference of NIHSS score between pre-treatment and at 72 hours (+/- 8 hours) after onset | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Shinichi Yoshimura, MD, PhD, Principal Investigator — Hyogo Medical University
Locations (1):
- Hyogo College of Medicine, Nishinomiya, Hyōgo, Japan

REFERENCES:
- [Derived] Roaldsen MB, Jusufovic M, Berge E, Lindekleiv H. Endovascular thrombectomy and intra-arterial interventions for acute ischaemic stroke. Cochrane Database Syst Rev. 2021 Jun 14;6(6):CD007574. doi: 10.1002/14651858.CD007574.pub3. PMID 34125952